CLINICAL TRIAL: NCT04288752
Title: CI03: A Clinical Investigation to Evaluate Efficacy of the J3 Bioscience Lubricating Intravaginal Ring VR101 as a Personal Lubricant Device in Women
Brief Title: Efficacy of VR101 as a Personal Lubricant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J3 Bioscience, Inc. (Industry)
Collaborators: Advanced Clinical Research Services, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CI03
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Sexual Dysfunction, Physiological
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, sham-controlled, 4-week parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double-blind, meaning the subject and Investigator/staff will not have access to or knowledge of the subject's treatment assignment. Further, since the Sponsor will securely maintain the randomization schedules, the Sponsor and Sponsor's representatives will not be made aware of a given subject's randomization arm until the blind is broken. The Sponsor will ensure that the Study Monitor does not ever have access to the randomization assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VR101 Lubricating Intravaginal Ring (Experimental): VR101 is a clear, flexible, torus-shaped lubricating intravaginal ring (IVR) manufactured from hollow tubing formed from Excipient Grade Thermoplastic Urethane Pathway® Polymer PY-PT42DE35 by hot-melt extrusion. Subjects randomized to this arm will be asked to use each ring for 7 days and replace with a new ring each week for 4 weeks. This will be followed by an optional 2-week open-label extension with active rings and a 1-week follow-up.
  Interventions: Device: VR101 Lubricating Intravaginal Ring
- Sham Ring (Sham Comparator): Performance of VR101 will be compared to that of an inactive ring. Subjects randomized to this arm will be asked to use each ring for 7 days and replace with a new ring each week for 4 weeks. This will be followed by an optional 2-week open-label extension with active rings and a 1-week follow-up.
  Sham rings are visually identical to VR101 Lubricating Intravaginal Rings, but no lubricating solution was added.
  Interventions: Device: Sham Ring

INTERVENTIONS:
Device: VR101 Lubricating Intravaginal Ring — VR101 Lubricating Intravaginal Ring is a personal lubrication device, for vaginal application, intended to moisturize and lubricate, to enhance the ease and comfort of intimate sexual activity, and supplement the body's natural lubrication.
  Other Names: Lubricating intravaginal ring
  Arms: VR101 Lubricating Intravaginal Ring
Device: Sham Ring — Sham rings are visually identical to VR101 Lubricating Intravaginal Rings, but no lubricating solution was added.
  Arms: Sham Ring

SUMMARY:
This Clinical Investigation (CI03) is designed to validate the efficacy of the VR101 lubricating Intravaginal Ring (IVR) as a personal lubricant device. In the proposed clinical investigation, participants will be randomized into two groups for the study, VR101 Active Ring and Inactive Ring. Participants will use VR101 active rings or inactive rings for 28 days in a randomized, double-blind, parallel group design. The study also includes an optional two-week open-label extension with active rings, and a one-week follow-up.

DETAILED DESCRIPTION:
BACKGROUND This study will look at the use of a study device that is intended to provide moisture and lubrication to enhance the ease and comfort of intimate sexual activity and supplement the body's natural lubrication. To date, regarding human clinical testing, the study device has been tested and evaluated in a human study with 72 female subjects and another study with 21 female subjects.

The purpose of this research study is to assess how safe and effective the study device (a vaginal ring referred to as VR101) is at providing personal lubrication. The study will compare the effectiveness of VR101 active ring compared to VR101 inactive ring, to enhance the ease and comfort of intimate sexual activity and supplement the body's natural lubrication. This is a research study to test a new investigational device. An investigational device is one that is not approved by the United States Food and Drug Administration (FDA). The study device is in the form of a clear, flexible ring that is placed in the vagina. Each ring is about 2 inches in diameter, or across the ring, from one side to the other.

During the study, participants will receive either the VR101 active ring or a ring that looks exactly like the VR101 ring but is inactive. For the purposes of this document, both VR101 active ring and the inactive ring will be referred to as the study ring, or study device.

Because this is a research study, study rings will be given to participants only during this study and must only be used according to the schedule that will be described by study staff. Participants will not be allowed to use them once the study is complete.

The results will be reported in a submission to the FDA to determine if the VR101 study device can be legally marketed in the United States.

PROCEDURES

Before any study-related tests and procedures are performed all subjects will read, sign, and date the consent document. Information will be collected after the consent document is signed and dated to determine eligibility to enroll in the study. This information includes demographic background, health, medical and social history, birth control method, prescribed medications, herbal or over the-counter drugs, use nonprescription drugs and alcohol. Women who are able to become pregnant will provide a urine sample for a pregnancy test. Potentially eligible subjects will complete the Female Sexual Function Index (FSFI) to assess sexual function in women who are sexually active. If all inclusion and exclusion criteria are satisfied, subjects will be enrolled and randomly assigned to the VR101 Active Ring or Inactive Ring treatment arm of the study.

About 160 female subjects will participate in this study. Upon meeting all inclusion/exclusion criteria, subjects will be randomized (1:1) to one of the two treatment arms and given a 4 week supply of the randomly assigned study devices. They will be instructed on how to use the ring and how to replace the ring weekly. During the 4-week treatment period, subjects will receive weekly phone calls to ensure compliance and collect information about sexual activity, ring replacement, and experience with the device. At the end of four weeks, each subject will return to the study site to complete the final study measures. They will return all unused study devices and undergo a urine sample pregnancy test if appropriate. They will complete the (FSFI) to assess the effects of the study device on sexual function after 4 weeks, and any changes to medications and health will be documented. At that time all subjects will be given the option of receiving an additional 2 weeks of the active VR101 study device.

ELIGIBILITY:
Inclusion Criteria: Clinical Investigation Participants Must:

1. Completely understand and sign the informed consent form (ability to read and understand the consent form in the English language).
2. Be at least 21 years of age.
3. Express a willingness to comply with the entire study visit schedule outlined in the protocol.
4. Over the course of the study:

   1. Abstain from the use of any vaginal moisturizers or lubricants or any other topically applied vaginal products not provided by study staff during the entirety of study participation
   2. Abstain from using lubricated or spermicide-containing male or female condoms
   3. Abstain from vaginal intercourse with a male partner using a lubricated condom
   4. Abstain from any oral sex during or prior to vaginal intercourse with a male partner.
   5. Must not initiate, modify or discontinue a regimen of HRT (hormone replacement therapy) or estrogen-containing birth control.

      NOTE: Women who have been using non-vaginal HRT or estrogen-containing birth control (e.g., oral, transdermal) on a regular dosing interval continuously for at least 3 months may continue on the same regimen during the study
   6. Abstain from the use of any other vaginally-placed devices (e.g. ring, diaphragm, cervical cap, pessary products)
   7. If able to get pregnant, use an approved method of contraception (per the remainder of I/E criteria) to reduce their risk of becoming pregnant during the study.
5. In the previous 3 months, have had or attempted sexual intercourse with a male partner a minimum of twice per month (on average).
6. Respond to all 4 individual FSFI Lubrication Questions (7 - 10) with a score of 1, 2, or 3.
7. Attempt sexual intercourse at least 4 times during the 4-week double-blind study.

Exclusion criteria for participant selection

Participants self-reporting any of the following will be ineligible for study entry:

1. Current use of HRT (Hormone Replacement Therapy) or any estrogen-containing birth control products, unless not applied vaginally and the participant has been on a regular dosing interval for at least 3 months prior and is willing to continue the same regimen without modification throughout study participation.
2. Vulvar or vaginal procedures (biopsies, radiation) in the last 3 months.
3. Active vulvar or vaginal infections/lesions or complaints, as well as undiagnosed abnormal genital bleeding.
4. History of chronic pelvic pain, interstitial cystitis, vulvar vestibulitis, pelvic inflammatory disease within the past 3 months.
5. Known current cervical or vaginal infection.
6. Participants who have given birth or terminated pregnancy in the past 6 weeks.
7. Postpartum or post-abortion endometritis, unless symptoms resolved at least 3 months prior to study entry.
8. Current persistent, abnormal vaginal bleeding.
9. History of the inability to place a vaginal ring.
10. History of any abnormality of the vagina resulting in distortion of the vaginal canal or incompatibility with vaginal ring placement.
11. Body habitus or history of lower genital tract abnormalities or prior surgeries, which may not allow the vagina to be appropriately accessed.
12. Known or suspected allergy or hypersensitivity to polyurethanes or glycerol.
13. Known current alcohol or illicit drug abuse.
14. Participants who have not recovered from adverse events due to chemotherapy or radiation treatment for cancer.
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection of the urogenital tract, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
16. Any condition that in the opinion of the investigator or study staff that would constitute contraindications to participation in the study or would compromise the ability to comply with the study protocol.
17. Current use of a vaginally-placed device (e.g., ring, pessary, cervical cap or diaphragm) unless willingness to discontinue for the study duration is expressed.
18. Pregnancy or plans to become pregnant in the next 6 months.
19. Current breastfeeding.
20. Participation in a previous ViroPan or J3 Bioscience clinical trial for VR101 (i.e., CI01, CI02)

NOTE: IUD (Intrauterine Device) users may be enrolled provided they commit to exercising caution when removing VR101, as IUD strings have been noted to interfere with VR101 removal.

NOTE: Participants who have previously undergone anterior and/or posterior vaginal repair and have received a vaginal mesh implant may have difficulty placing VR101 but are not automatically excluded from the study.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler McCabe, PhD, Study Director — J3 Bioscience, Inc.
Locations (2):
- United States (2):
  - Advanced Clinical Research, Inc. (ACR Idaho), Meridian, Idaho
  - Advanced Clinical Research, Inc. (ACR Utah), West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: None. Each enrolled subject was randomly assigned in a 1:1 ratio to receive either VR101 devices or sham rings. One enrolled subject was randomized but did not begin the treatment phase because she was unable to place the first device.
Period: Overall Study
Arm/Group | VR101 Lubricating Intravaginal Ring | Sham Ring
Started | 87 (88 Participants were randomized to the VR101 group. However, one randomized participant (AR33) was unable to place the device and was immediately terminated from the study, prior to any post-randomization data collection. Therefore, 87 participants assigned to the VR101 group entered the treatment phase.) | 88
Completed | 81 | 85
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Sham Ring: Performance of VR101 will be compared to that of an inactive ring. Subjects randomized to this arm will be asked to use each ring for 7 days and replace with a new ring each week for 4 weeks. This will be followed by an optional 2-week open-label extension with active rings and a 1-week follow-up.
  Sham rings are visually identical to VR101 Lubricating Intravaginal Rings, but no lubricating solution was added.
  Sham Ring: Sham rings are visually identical to VR101 Lubricating Intravaginal Rings, but no lubricating solution was added.
- Total: Total of all reporting groups
Arm/Group | VR101 Lubricating Intravaginal Ring | Sham Ring | Total
Number analyzed (Participants) | 87 | 88 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.4) | 47.1 (13.0) | 49.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 88 | 175
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 81 | 83 | 164
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  White | 86 | 84 | 170
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Increased Female Sexual Function Index Lubrication Domain (FSFI-LD) Scores
Description: The Female Sexual Function Index (FSFI) is a survey validated to assess sexual function in women. The FSFI contains 19 questions, divided in to 6 characteristic domains: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. Although all of these characteristics may be improved by use of a personal lubricant, only the Lubrication Domain (FSFI-LD) is directly relevant to a lubricant's intended use.
  Primary Endpoint: Proportion of participants that experience increased vaginal lubrication that enhances ease and comfort of intimate sexual activity, defined as an FSFI-LD ≥ 4.5 (out of 6.0) with 4 consecutive weeks of weekly ring use.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VR101 Lubricating Intravaginal Ring | Sham Ring
Number analyzed (Participants) | 87 | 88
Participants | 57 | 43

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 5-7 weeks per participant.
Arm/Group | VR101 Lubricating Intravaginal Ring | Sham Ring
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/88
Other Adverse Events (participants affected / at risk) | 36/87 | 26/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VR101 Lubricating Intravaginal Ring (N=87) | Sham Ring (N=88)
Excess Vaginal Secretions / Lubrication / Discharge - Moderate (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Excess Vaginal Secretions / Lubrication / Discharge - Mild (Reproductive system and breast disorders) | 10 (11) | 2 (2)
Pelvic / Reproductive Tract Cramping - Moderate (Reproductive system and breast disorders) | 2 (3) | 1 (1)
Pelvic / Reproductive Tract Cramping (Reproductive system and breast disorders) | 8 (8) | 2 (2)
Vaginal Pain / Discomfort - Moderate (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Pain / Discomfort - Mild (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Non-Menstrual Bleeding (Reproductive Tract) - Moderate (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Non-Menstrual Bleeding (Reproductive Tract) - Mild (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Increased Urinary Urge / Urinary Incontience - Moderate (Renal and urinary disorders) | 1 (1) | 0 (0)
Increased Urinary Urge / Urinary Incontience - Mild (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary Tract / Bladder Infection - Moderate (Renal and urinary disorders) | 2 (2) | 1 (1)
Vaginal Irritation / Vaginitis - Moderate (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal Yeast Infection - Mild (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Device Interference with Intercourse - Mild (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile Discomfort (Partner) - Mild (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hot Flashes - Mild (General disorders) | 1 (1) | 0 (0)
Burning During Urination - Mild (Renal and urinary disorders) | 1 | 0 (0)
Intermittent Headaches - Mild (General disorders) | 1 (1) | 0 (0)
Abdominal Cramping - Mild (General disorders) | 0 (0) | 1 (1)
Nausea - Mild (General disorders) | 0 (0) | 1 (1)
Bladder Spasms - Mild (Renal and urinary disorders) | 0 (0) | 1 (1)
Other - Not Related to Device (General disorders) | 12 (13) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT04288752/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT04288752/SAP_001.pdf